CLINICAL TRIAL: NCT06879626
Title: Effect of Pecan Consumption on Aging
Brief Title: Effect of Snacks on Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: American Pecan Promotion Board (Unknown)
Responsible Party: Principal Investigator, Zhaoping Li, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-25-0037
Record Dates: First submitted 2025-02-11; First posted 2025-03-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pecan arm (Experimental): Participats in this arm will be comsuming 2 oz of pecans daily for 12 wekks
  Interventions: Other: Pecan
- Pretzel arm (Experimental): Participants in this arm will consume 3.5 oz of pretzel snacks daily for 12 weeks
  Interventions: Other: Pretzel

INTERVENTIONS:
Other: Pecan — 2 oz of whole raw pecans
  Arms: Pecan arm
Other: Pretzel — 3.5 oz of pretzel snacks daily
  Arms: Pretzel arm

SUMMARY:
The purpose of this study is to determine if daily consumption of 2 oz of pecans compared to 3.5 oz pretzel snacks for 12 weeks will 1) contribute to the body's ability to protect itself from oxidative damage (caused by oxygen radicals created by ultraviolet (UV) B light) by evaluating skin resistance to UV light irritation, skin fats/oils degradation and "rusting", and oxidative damage to the skin genes; and 2) explore the mechanisms of how snack consumption may affect aging by analyzing blood markers of aging as well as the microbes living in the gut (gut microbiome).

DETAILED DESCRIPTION:
Oxidative stress plays a significant role in the aging process. Antioxidant potential of tree nuts, including pecans, has been previously reported. However, very few studies have evaluated the antioxidant effects and their underlying mechanisms of nut consumption in the aging population. Skin is the largest organ and is the first body part to exhibit signs of aging. Human skin exposed to solar ultraviolet radiation (UVR) experiences a dramatic increase in production of reactive oxygen species (ROS) and inflammation. Moreover, skin aging is associated with increased levels of oxidative stress. Investigators previously showed that almond and pomegranate consumption can improve the antioxidant defense of skin by reducing UV-induced damage. In addition, the prebiotic properties of nuts and other bioactive-rich foods have been of great interest lately, current study team and others have reported the gut microbiome modulating effects of tree nut consumption. Based on this evidence and other published data, it is being proposed that pecans, due to their bioactive compound content, may have the potential to contribute to whole body antioxidant protection, modulate the gut microbiome and affect the aging process. The aim of this study is to evaluate the effects of incorporating 2 oz of pecans into diet compared to isocaloric pretzel snacks daily for 12 weeks 1) on whole body antioxidant capacity by evaluating skin resistance to UV irritation, lipid oxidation, and oxidative DNA damage; and 2) explore the mechanism of how pecan consumption affects aging by analyzing circulating biomarkers of aging as well as the gut microbiome. This will be a two-arm, randomized, placebo-controlled intervention study in 60 middle-aged and older generally healthy non-vegetarian/vegan women (age 55-75 years, Fitzpatrick's skin types II-IV). Investigating the effects of pecan consumption on skin antioxidant defense and systemic oxidative status will uncover valuable new insights into whether bioactive compounds in pecans can contribute to the total body antioxidant capacity and affect the aging process.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Generally healthy
* Aged 55-75 years
* BMI 18.5-34.9 kg/m2
* Fitzpatrick Skin type II-IV
* Consume a typical Western diet (low in polyphenols-rich foods and fiber)
* Willing to maintain habitual dietary and exercise patterns for the study duration
* Willing to maintain normal skin care products and pattern for the duration of the study
* Willing to come to study visits without any makeup and skin products on
* Subjects must read and sign the Institutional Review Board-approved written informed consent prior to the initiation of any study specific procedures or enrollment. A subject will be excluded for any condition that might compromise the ability to give truly informed consent.

Exclusion Criteria:

* Vegetarian/vegan
* Known nut allergy
* Skin-related prescription medication, supplements or non-prescription cosmeceutical agents
* Initiation of topical or oral prescription steroids and/or anti-inflammatory medications within 30 days prior to study enrollment
* Excessive exposure to either natural or artificial sunlight
* Screening laboratory values outside of the normal range that is considered clinically significant for study participation by the investigator
* Documented chronic disease
* Taking medications or supplements known to affect gut microbiota composition (antibiotics within the past 3 months, probiotics, fiber, etc.)
* Taking exogenous hormones (e.g. hormone replacement therapy)
* Recent weight fluctuations (>10% in the last 6 months)
* Smoker or living with a smoker
* Use of >20 g of alcohol per day
* Unable or unwilling to comply with the study protocol (including unwillingness to avoid nuts for the whole duration of the study)
* Unable to provide consent
* Pregnancy and/or lactation

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Minimal Erythema Dose (MED) | At baseline and 12 weeks
  To determine the minimal erythema dose (MED) at the inner arm, skin UVB dose and treatment time will be determined based on overall skin type classification. Based on overall skin type classification we will use the National Biological UVB mJ chart to determine the dose and sequential exposure times for each skin patch. A sleeve with 6 cutout patches will be placed on participant's arm. Using the Dermalight 90 handheld device (National Biological, Beachwood, OH) each cutout test area on the inner arm of subjects will be exposed to a defined dose of narrow band ultraviolet B (NB-UVB) light delivered by the UV exposure between 270 and 400 nm. Each cutout window will be exposed to an increasing dose. To evaluate the minimal erythema dose (MED) participants will need to return 24 hours later to determine which skin patch showed minimal erythema (pink color). Although 6 cutouts will be made, this is a single outcome measure as the all 6 cutouts will all be measuring MED in mJ/cm^2.

SECONDARY OUTCOMES:
Skin characteristics | At baseline and 12 weeks
  skin elasticity (Cutometer Dual MPA 580) in N/m
Skin characteristics | At baseline and 12 weeks
  hydration (Corneometer CM 825) in AU
Skin characteristics | At baseline and 12 weeks
  color (Mexameter MX18) in AU
Skin characteristics | At baseline and 12 weeks
  skin gloss (SkinGlossymeter GL200) in GU

OTHER OUTCOMES:
Biomarkers of aging and inflammation | At baseline and 12 weeks
  C-C motif chemokine 27 (CTACK/CCL27) in pg/ml
Biomarkers of aging and inflammation | At baseline and 12 weeks
  fibroblast growth factor 21 (FGF-21) in pg/ml
Biomarkers of aging and inflammation | At baseline and 12 weeks
  growth/differentiation factor 11 (GDF-11) in ng/ml
Biomarkers of aging and inflammation | At baseline and 12 weeks
  growth/differentiation factor 15 (GDF-15) in pg/ml
Biomarkers of aging and inflammation | At baseline and 12 weeks
  gonadoliberin (GnRH) in pg/ml
Biomarkers of aging and inflammation | At baseline and 12 weeks
  interleukin-6 (IL-6) in pg/ml
Biomarkers of aging and inflammation | At baseline and 12 weeks
  interleukin-10 (IL-10) in pg/ml
Biomarkers of aging and inflammation | At baseline and 12 weeks
  interleukin-18 (IL-18) in pg/ml
Biomarkers of aging and inflammation | At baseline and 12 weeks
  Jagged 1 protein (Jag1) in kDA
Biomarkers of aging and inflammation | At baseline and 12 weeks
  leptin in ng/ml
Oxidative stress markers | At baseline and 12 weeks
  Urine malondialdehyde (MDA) in ng/ml
Oxidative stress markers | At baseline and 12 weeks
  Blood MDA in nmol/ml
Oxidative stress markers | At baseline and 12 weeks
  Urine 8OHdG in ng/mg creatinine
Oxidative stress markers | At baseline and 12 weeks
  Blood 8OHdG in ng/ml
Gut microbiome | At baseline and 12 weeks
  The stool specimen will be collected by the participants at home at baseline and week 12 utilizing our Stool Collection Kit as per instructions. Immediately after collection, the specimen will be frozen in a home freezer and delivered in an insulated container to the UCLA Center for Human Nutrition. At UCLA, the specimen will be stored at - 80 ºC. Fecal microbiological analyses. Approximately 1g of the stool will be weighed and dried in a vacuum drying oven (15 in Hg) at 80 ºC for 48 hours, then weighed again to establish the moisture content so that all counts can be corrected to dry weight. From another aliquot of remaining fecal samples, DNA will be extracted using bead beating with a commercial extraction system (DNeasy PowerSoil® DNA Isolation Kit, Qiagen, Valencia, CA). The quality of the DNA samples will be confirmed using a Nanodrop 1000 (Thermo Fisher Scientific, Wilmington, DE). Extracted DNA will be transferred to UCLA Microbiome Core facility for MiSeq sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Center for Human Nutrition, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
Data analysis will be performed in-house.